CLINICAL TRIAL: NCT02032875
Title: A Phase 3 Evaluation of Daclatasvir, Sofosbuvir, and Ribavirin in Genotype 1-6 Chronic Hepatitis C Infection Subjects With Cirrhosis Who May Require Future Liver Transplant and Subjects Post-Liver Transplant
Brief Title: Phase III Daclatasvir, Sofosbuvir, and Ribavirin in Cirrhotic Participants and Participants Post-liver Transplant
Acronym: ALLY 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-215
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-liver Transplant Cohort (Experimental): Participants with liver transplant received daclatasvir 60 mg, sofosbuvir 400 mg, and ribavirin (based on baseline hemoglobin and creatinine clearance and tolerated dose) tablets daily for 12 weeks and were followed for 24 weeks post treatment.
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir; Drug: Ribavirin
- Cirrhotic Cohort (Experimental): Cirrhotic participants received daclatasvir 60 mg, sofosbuvir 400 mg, and ribavirin (based on baseline hemoglobin and creatinine clearance and tolerated dose) tablets orally for 12 weeks and were followed for 24 weeks post-treatment. Cirrhotic participants who received a liver transplant while on study treatment were eligible (>3 months post transplant) for a treatment extension of daclatasvir 60 mg, sofosbuvir 400 mg, and ribavirin (dose based on hemoglobin level) tablets orally for an additional 12 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Sofosbuvir
Drug: Ribavirin

SUMMARY:
This trial was open to participants who had received a liver transplant or had cirrhosis due to chronic HCV. All subjects were treated with daclatasvir+sofosbuvir+ribavirin and were followed for 24 weeks post treatment. Under certain conditions, the treatment duration could have been extended for cirrhotic participants. The study tested the efficacy and safety of this combination for treatment of HCV in cirrhotic and post transplant patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must be able to understand and agree to comply with the prescribed dosing regimens and procedures, report for regularly scheduled study visits, and reliably communicate with study personnel about adverse events and concomitant medications
* Participants chronically infected with hepatitis C virus (HCV) Genotype 1, 2, 3, 4, 5, or 6 with HCV RNA viral load of ≥10,000 IU/mL at screening
* Participants may be treatment-naïve or treatment-experienced
* Cirrhotic participants must have cirrhosis confirmed by biopsy, Fibroscan or fibrotest and Aspartate aminotransferase platelet ratio index (APRI) criteria as outlined in the protocol
* Post-transplant participants must be at least 3 months post-transplant with no evidence of moderate or severe rejection

Exclusion Criteria:

* History of multi-organ transplant, with the exception of dual transplantation of the liver/kidney, is prohibited
* Current or known history of cancer (with the following exceptions: In situ carcinoma of the cervix, adequately treated basal or squamous cell carcinoma of the skin, or hepatocellular carcinoma within Milan criteria for transplantation) within 5 years prior to screening
* Evidence of an ongoing medical condition contributing to chronic liver disease other than HCV (such as, but not limited to: hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, or toxin exposures)
* History of HIV infection or chronic hepatitis B virus (HBV) as documented by HBV serologies (e.g., HBsAg-seropositive). Participants with resolved HBV infection may participate (e.g., HBcAb-seropositive with concurrent HBsAg-seronegative)
* Active hospitalization for decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - University Of Miami Schiff Center For Liver Diseases, Miami, Florida
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Baylor St. Luke'S Medical Center, Houston, Texas
  - American Research Corporation, San Antonio, Texas
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 centers in the United States.
Pre-assignment Details: A total of 116 participants were enrolled, of which 113 received study treatment (60 cirrhotic cohort, 53: post-liver transplant cohort). Remaining 3 participants no longer met study criteria. Of the 60 participants in the cirrhotic cohort, 57 did not receive a treatment extension and 3 received a treatment extension after liver transplant.
Groups:
- Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin: Participants with liver transplant, received 12 weeks of daclatasvir 60-mg and sofosbuvir 400-mg once daily (QD) orally, with ribavirin at a recommended initial dose of 600 mg and were followed for 24 weeks post-treatment. The dose of ribavirin could be titrated to 1000 mg/day if tolerated.
- Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin: Participants received 12 weeks of daclatasvir 60-mg and sofosbuvir 400-mg once daily (QD) orally, with ribavirin at a recommended initial dose of 600 mg and were followed for 24 weeks post-treatment. The dose of ribavirin could be titrated to 1000 mg/day if tolerated.
Period: Treatment Period
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Started | 53 | 60
Completed | 52 | 56
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Liver transplant, No extension needed | 0 | 1
Not completed — Liver transplant, Treatment extension | 0 | 3
Period: Follow-up Period
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Started | 53 (Out of 53 participants who entered the treatment period, all 53 continued in the follow-up period.) | 57 (Of 60 participants in treatment period, 57 continued in follow-up, 3 entered treatment extension.)
Completed | 50 | 46
Not Completed | 3 | 11
Not completed — Death | 0 | 1
Not completed — Virologic Relapse | 3 | 10

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of active study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Total
Number analyzed (Participants) | 53 | 60 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.25) | 57.9 (9.45) | 58.7 (8.91)
Age, Customized [Number; unit: participants]
  <65 years | 42 | 50 | 92
  >=65 years | 11 | 10 | 21
Gender [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 38 | 38 | 76
Hepatitis C Virus RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.61 (0.711) | 6.01 (0.617) | 6.29 (0.724)
Hepatitis C Virus RNA distribution [Number; unit: participants]
  <800,000 IU/mL | 6 | 27 | 33
  ≥800,000 IU/mL | 47 | 33 | 80
HCV genotype subtype [Number; unit: participants]
  Hepatitis C Virus genotype 1a | 31 | 34 | 65
  Hepatitis C Virus genotype 1b | 10 | 11 | 21
  Hepatitis C Virus genotype 2 | 0 | 5 | 5
  Hepatitis C Virus genotype 3 | 11 | 6 | 17
  Hepatitis C Virus genotype 4 | 0 | 4 | 4
  Hepatitis C Virus genotype 5 | 0 | 0 | 0
  Hepatitis C Virus genotype 6 | 1 | 0 | 1
IL-28B rs1297860 Genotype [Number; unit: participants]
  CC | 13 | 13 | 26
  CT | 31 | 33 | 64
  TT | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HCV Genotype-1 Infected Post-liver Transplanted Participants With Sustained Virologic Response at Post-treatment Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C Virus (HCV) RNA levels below the lower limit of quantitation (<LLOQ) i.e., 25 IU/mL target detected or target not detected, at post-treatment Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: Post-treatment follow-up Week 12
Population: All HCV genotype 1 infected post-transplant participants who received at least 1 dose of study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 41
Percentage of participants | 95.1 [83.5 to 99.4]

2. Primary Outcome: Percentage of Genotype-1 Infected Cirrhotic Participants With Sustained Virologic Response at Post-treatment Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C Virus (HCV) RNA levels below the lower limit of quantitation i.e., 25 IU/mL target detected or target not detected, at post-treatment Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: Post-treatment follow-up Week 12
Population: All genotype 1 cirrhotic participants who received at least 1 dose of study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 45
Percentage of participants | 82.2 [67.9 to 92.0]

3. Secondary Outcome: Percentage of Participants Who Achieved Sustained Virologic Response at Post-treatment Week 12 (SVR12) for All Genotypes and Genotypes 2, 3, 4, 6
Description: as for outcome 2
Time Frame: Post-treatment follow-up Week 12
Population: All treated participants who took at least 1 dose of study medication. Here, 'n' signifies participants evaluable for SVR12 at the specified time point in each group, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
Percentage of participants
  All Genotypes (n =53, 60) | 94.3 [84.3 to 98.8] | 83.3 [71.5 to 91.7]
  HCV Genotype 2 (n =0, 5) | NA [NA to NA] — As none of the participants were evaluable for this reporting arm, the percentage value was not applicable. | 80 [28.4 to 99.5]
  HCV Genotype 3 (n =11, 6) | 90.9 [58.7 to 99.8] | 83.3 [35.9 to 99.6]
  HCV Genotype 4 (n =0, 4) | NA [NA to NA] — As none of the participants were evaluable for this reporting arm, the percentage value was not applicable. | 100 [39.8 to 100]
  HCV Genotype 6 (n =1, 0) | 100 [2.5 to 100] | NA [NA to NA] — As none of the participants were evaluable for this reporting arm, the percentage value was not applicable.

4. Secondary Outcome: Percentage of Participants Who Achieve Hepatitis C Virus RNA Levels Below the Lower Limit of Quantitation Target Detected or Target Not Detected at Each of the Following Weeks: 1, 2, 4, 6, 8, 12, End of Treatment; Follow Up Weeks 4, 8, and 24
Description: Participants who responded to treatment were assessed using proportion of subjects with hepatitis C Virus RNA levels below the lower limit of quantitation i.e., 25 IU/mL target detected or target not detected, at each visit.
Time Frame: Week 1, 2, 4, 6, 8, 12, End of treatment, Follow-up Week 4, 8, and 24
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
Percentage of participants
  Week 1 | 22.6 [12.3 to 36.2] | 15.0 [7.1 to 26.6]
  Week 2 | 67.9 [53.7 to 80.1] | 45.0 [32.1 to 58.4]
  Week 4 | 94.3 [84.3 to 98.8] | 95.0 [86.1 to 99.0]
  Week 6 | 96.2 [87.0 to 99.5] | 91.7 [81.6 to 97.2]
  Week 8 | 98.1 [89.9 to 100] | 95.0 [86.1 to 99.0]
  Week 12 | 98.1 [89.9 to 100] | 93.3 [83.8 to 98.2]
  End of treatment | 100.0 [93.3 to 100.0] | 96.7 [88.5 to 99.6]
  Follow-up Week 4 (SVR4) | 98.1 [89.9 to 100] | 88.3 [77.4 to 95.2]
  Follow-up Week 8 (SVR8) | 96.2 [87 to 99.5] | 86.7 [75.4 to 94.1]
  Follow-up Week 24 (SVR24) | 94.3 [84.3 to 98.8] | 80.0 [67.7 to 89.2]

5. Secondary Outcome: Percentage of Participants Who Achieve Hepatitis C Virus RNA Levels Below the Lower Limit of Quantitation Target Not Detected at Each of the Following Weeks: 1, 2, 4, 6, 8, 12, End of Treatment
Description: Participants who responded to treatment were assessed using proportion of subjects with hepatitis C Virus RNA levels below the lower limit of quantitation i.e., 25 IU/mL target not detected, at each on-treatment visit.
Time Frame: Week 1, 2, 4, 6, 8, 12, End of treatment
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
Percentage of participants
  Week 1 | 3.8 [0.5 to 13.0] | 1.7 [0.0 to 8.9]
  Week 2 | 13.2 [5.5 to 25.3] | 11.7 [4.8 to 22.6]
  Week 4 | 56.6 [42.3 to 70.2] | 53.3 [40.0 to 66.3]
  Week 6 | 84.9 [72.4 to 93.3] | 76.7 [64.0 to 86.6]
  Week 8 | 98.1 [89.9 to 100] | 93.3 [83.8 to 98.2]
  Week 12 | 98.1 [89.9 to 100.0] | 93.3 [83.8 to 98.2]
  End of treatment | 100.0 [93.3 to 100.0] | 96.7 [88.5 to 99.6]

6. Secondary Outcome: Percentage of Participants With CC or Non-CC Genotype Who Achieved Sustained Virologic Response at 12 Weeks After the Last Dose of Study Drug (SVR12)
Description: Participants categorized into 2 genotypes (CC and non-CC) based on single nucleotide polymorphism in the IL28B gene were assessed for SVR12, defined as response in which hepatitis C virus RNA levels be <lower limit of quantitation ie, 25 IU/mL or below target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. For participants who missed the follow-up Week 12 visit, SVR12 was imputed using the next and closest available HCV RNA measurement after the follow-up Week 12 window.
Time Frame: Post-treatment follow-up Week 12
Population: All treated participants. Here, 'n' signifies participants evaluable for SVR12 at the specified time point in each group, respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
Percentage of participants
  CC type (n = 13, 13) | 100 [75.3 to 100] | 84.6 [54.6 to 98.1]
  Non-CC type (n = 40, 47) | 92.5 [79.6 to 98.4] | 78.7 [64.3 to 89.3]

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), AEs Leading to Interruption, Treatment-related AEs/SAEs, Grade 3 to 4 AEs/SAEs, and Death
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From start of study treatment up to 7 days post last dose of study treatment (approximately 13 weeks)
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
participants
  SAEs | 5 | 10
  AEs leading to discontinuation | 6 | 10
  AEs leading to interruption | 1 | 3
  Treatment-related AEs | 35 | 37
  Treatment-related SAEs | 0 | 0
  Adverse events Grade 3 to 4 | 5 | 11
  Serious adverse events Grade 3 to 4 | 2 | 8
  Death | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment Emergent Grade 3-4 Laboratory Abnormalities
Description: Grade 3-4 laboratory abnormalities were defined as: Hemoglobin as 6.50-7.4 g/dL for grade 3 and/or < 6.5 g/dL for grade 4, Platelet count as 25*10^9-50*10^9 /L for grade 3 and/or < 25.000*10^9 /L for grade 4, International normalized ratio as 2.1-3.0*upper limit of normal (ULN) > 3.0*ULN for grade 3 and/or > 3.0*ULN for grade 4, Leukocytes as 1.0*10^9-1.5*10^9/L for grade 3 and/or <1.0*10^9/L for grade 4, Lymphocytes (Absolute) as 0.350*109-0.499*10^9 /L for grade 3 and/or < 0.350*10^9 /L for grade 4, Alanine aminotransferase as 5.1-10.0*ULN for grade 3 and/or > 10.0*ULN for grade 4, Aspartate aminotransferase as 5.1-10.0*ULN for grade 3 and/or > 10.0*ULN for grade 4, Alkaline phosphatase as 5.1-10.0*ULN for grade 3 and/or > 10.0*ULN for grade 4, Bilirubin (Total) as 2.6-5.0*ULN for grade 3 and/or > 5.0*ULN for grade 4, Albumin as < 20 g/L, Lipase (Total) as 3.1-5.0*ULN for grade 3 and/or > 5.0*ULN for grade 4, and Creatinine as 1.9-3.4*ULN for grade 3 and/or ≥ 3.5*ULN for grade 4.
Time Frame: From start of study treatment up to 7 days post last dose of study treatment
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Number analyzed (Participants) | 53 | 60
participants
  Hemoglobin | 2 | 5
  Platelet count | 0 | 4
  International normalized ratio | 0 | 1
  Leukocytes | 2 | 0
  Lymphocytes (Absolute) | 3 | 6
  Alanine aminotransferase | 0 | 2
  Aspartate aminotransferase | 0 | 3
  Alkaline phosphatase | 1 | 0
  Bilirubin (Total) | 2 | 9
  Albumin | 0 | 1
  Lipase (Total) | 2 | 3
  Creatinine | 2 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 up to 7 days post last dose of study treatment (approximately 13 weeks)
Description: Study Start: March 17, 2014; Study Completion: January 5, 2016
Arm/Group | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin
Serious Adverse Events (participants affected / at risk) | 5/53 | 10/60
Other Adverse Events (participants affected / at risk) | 38/53 | 42/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin (N=53) | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin (N=60)
Encephalopathy (Nervous system disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post-liver Transplant Cohort: Daclatasvir+Sofosbuvir+Ribavirin (N=53) | Cirrhotic Cohort: Daclatasvir+Sofosbuvir+Ribavirin (N=60)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 10 | 5
Anaemia (Blood and lymphatic system disorders) | 11 | 13
Somnolence (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 19 | 9
Fatigue (General disorders) | 15 | 11
Oedema peripheral (General disorders) | 4 | 4
Dizziness (Nervous system disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 4 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Pyrexia (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.